CLINICAL TRIAL: NCT01314352
Title: A Randomized, Single-Dose, Two-Way Crossover Relative Bioavailability Study of Desloratadine 5 mg Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Bioavailability Study of Desloratadine 5 mg Tablet of Dr. Reddy's Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. M.S. Mohan/Vice President - R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 50486
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desloratadine Tablets, 5 mg (Experimental): Desloratadine Tablets, 5 mg of Dr. Reddy's Laboratories
  Interventions: Drug: Desloratadine
- Clarinex (Active Comparator): Clarinex® 5 mg Tablets of Schering-Plough
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — Desloratadine Tablets, 5 mg
  Other Names: Clarinex® 5 mg

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of Dr. Reddy's Desloratadine 5 mg tablet to that of Clarinex® 5 mg tablet in healthy subjects under fed conditions.

DETAILED DESCRIPTION:
A Randomized, Single-Dose, Two-Way Crossover Relative Bioavailability Study of Desloratadine 5 mg Tablet in fed Normal,Healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Is the individual a healthy, normal adult man and women who volunteers to participate?
* Is s/he within 18 and 45 years of age, inclusive?
* Is his/her BMI between 19 and 30, inclusive?
* Is she willing to avoid pregnancy by abstaining from sexual intercourse with a non-sterile male partner, or by the use one of the following methods: diaphragm + spermicide or condom + spermicide (at least 14 days before dosing), intra-uterine contraceptive device or hormonal contraceptives (at least 4 weeks prior to dosing), or has she been surgically sterile or post-menopausal at least six months prior to entering into the study?
* Is s/he considered reliable and capable of understanding his/her responsibility and role in the study?
* Has s/he provided written informed consent?

A no answer to any of the above questions indicates that the individual is ineligible for enrollment

Exclusion Criteria:

Does the individual have a history of allergy or hypersensitivity to desloratadine?

* Does s/he have clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Does s/he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, or renal diseases that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Is she nursing?
* Does s/he have serious psychological illness?
* Does s/he have significant history (within the past year) or clinical evidence of alcohol or drug abuse?
* Does s/he have a positive urine drug screen or a positive HIV-1, or hepatitis B or C screen, or a positive pregnancy test?
* Is s/he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 48 hours prior to study drug administration and ending when the last blood sample has been taken in each study period? .
* Has s/he used any prescription drug, other than hormonal contraceptives, during the 14-day period prior to study initiation, or any OTC drug during the 72-hour period preceding study initiation?
* Is s/he unable to refrain from the use of all concomitant medications, other than hormonal contraceptives, during the study?
* Has s/he donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation?
* Has s/he donated plasma during the two week period preceding study initiation?
* Has s/he used any tobacco products in the 3 months preceding drug administration?
* Has s/he received an investigational drug during the 30 day period preceding study initiation? A yes answer to any of the above questions indicates that the individual is ineligible for enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2005-12; Primary Completion 2005-12 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability is based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R. Pizarro, M.D.,, Principal Investigator — SFBC Ft. Myers, Inc
Locations (1):
- SFBC, Ft. Myers, Inc.,, Fort Myers, Florida, United States